CLINICAL TRIAL: NCT05229900
Title: A Phase 1 Study of SGN-ALPV in Advanced Solid Tumors
Brief Title: A Study of SGN-ALPV in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed due to portfolio prioritization
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGNALPV-001
Record Dates: First submitted 2022-01-26; First posted 2022-02-08 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Neoplasms; Endometrial Neoplasms; Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Gastroesophageal Junction Carcinoma; Uterine Cervical Neoplasms; Testicular Neoplasms
Keywords: Ovarian cancer; Endometrial cancer; Non-small cell lung cancer; NSCLC; Gastric cancer; GEJ carcinoma; Cervical cancer; Malignant Testicular Germ Cell Tumor; Malignant Ovarian Germ Cell Tumor; Malignant Extragonadal Germ Cell Tumor; High-grade serous ovarian cancer; HGSOC; Seattle Genetics
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Uterine Cervical Neoplasms; Testicular Neoplasms; Ovarian Germ Cell Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SGN-ALPV (Experimental): SGN-ALPV monotherapy
  Interventions: Drug: SGN-ALPV

INTERVENTIONS:
Drug: SGN-ALPV — Given into the vein (IV; intravenously)

SUMMARY:
This study will test the safety of a drug called SGN-ALPV in participants with solid tumors. It will also study the side effects of this drug. A side effect is anything a drug does to your body besides treating your disease.

Participants will have solid tumor cancer that has spread through the body (metastatic) or cannot be removed with surgery (unresectable).

This study will have three parts. Parts A and B of the study will find out how much SGN-ALPV should be given to participants. Part C will use the dose and schedule found in Parts A and B to find out how safe SGN-ALPV is and if it works to treat solid tumor cancers.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have one of the following histologically or cytologically confirmed metastatic or unresectable solid tumor types:

  * Parts A and B

    * Ovarian cancer
    * Endometrial cancer
    * Non-small cell lung cancer (NSCLC)
    * Gastric cancer, including gastroesophageal junction (GEJ) carcinoma
    * Cervical cancer
    * Malignant testicular germ cell tumor (GCT), except for pure teratomas
    * Malignant ovarian GCT, except for pure teratomas
    * Malignant extragonadal GCT except for pure teratomas or tumors with primaries arising from CNS
  * Part C

    * High-grade serous ovarian cancer (HGSOC): Participants must have HGSOC which has progressed or relapsed within 6 months after previous platinum containing chemotherapy, received 2 to 4 prior anticancer lines of therapy, and at least 1 line of therapy in the platinum-resistant setting. If eligible at least 1 line of therapy must have contained bevacizumab or a biosimilar to bevacizumab.
    * Endometrial Cancer: Participants must have unresectable locally advance or metastatic endometrial carcinoma and have had at least 1 prior line of therapy.
    * NSCLC: Participants must have unresectable locally advanced or metastatic NSCLC and have received platinum-based therapy and a PD-(L)1 inhibitor.
    * Gastric cancer or GEJ carcinoma: Participants must have unresectable locally advanced or metastatic gastric cancer or GEJ carcinoma and have received prior platinum and fluoropyrimidine -based chemotherapy
* Participants enrolled in the following study parts should have an appropriate tumor site and agree to a biopsy

  * Part B dose and schedule optimization cohorts and Part C disease-specific expansion cohorts: pretreatment biopsy, unless clinically infeasible following consultation with the medical monitor.
  * Part C biology expansion cohort: pretreatment biopsy (required), on-treatment biopsy during Cycle 1 (unless clinically infeasible following consultation with the medical monitor)
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Measurable disease per the RECIST v1.1 at baseline

Exclusion Criteria:

* History of another malignancy within 3 years of first dose of study treatment or any evidence of residual disease from a previously diagnosed malignancy. Exceptions are malignancies with a negligible risk of metastasis or death.
* Known active central nervous system metastases.
* Previous receipt of an MMAE-containing agent or an agent targeting ALPP or ALPPL2.
* Pre-existing neuropathy ≥ Grade 2 per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Through 30-37 days after last study treatment, approximately 6 months
  Any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Number of participants with laboratory abnormalities | Through 30-37 days after last study treatment, approximately 6 months
Number of participants with dose-limiting toxicities (DLTs) | Up to 28 days
Number of participants with DLTs by dose level | Up to 28 days

SECONDARY OUTCOMES:
Incidence of antidrug antibodies (ADAs) | Through 30-37 days after last study treatment, approximately 6 months
Area under the concentration-time curve (AUC) | Through 14 days after last study treatment, approximately 6 months
  PK parameter
Maximum concentration (Cmax) | Through 14 days after last study treatment, approximately 6 months
  PK parameter
Time to Cmax (Tmax) | Through 14 days after last study treatment, approximately 6 months
  PK parameter
Apparent terminal half-life (t1/2) | Through 14 days after last study treatment, approximately 6 months
  PK parameter
Trough concentration (Ctrough) | Through 14 days after last study treatment, approximately 6 months
  PK parameter
Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | Approximately 2 years
  The proportion of participants with an objective response (OR) per investigator. A participant is determined to have an OR if, based on RECIST v1.1, the subject achieves a complete response (CR) or a partial response (PR) after initiation of treatment and at or prior to the end of treatment (EOT) disease assessment.
Duration of objective response (DOR) | Approximately 2 years
  The time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of disease progression (based on radiographic assessments per RECIST v1.1) or death due to any cause.
Progression-free survival (PFS) | Approximately 2 years
  The time from start of study treatment to first documentation of disease progression or death due to any cause
Overall survival (OS) | Approximately 2 years
  The time from start of study treatment to death due to any cause
CA-125 response rate according to Gynecological Cancer Intergroup (GCIG) criteria (subjects with ovarian cancer only) | Approximately 2 years
  The proportion of participants with ovarian cancer who have at least a 50% reduction in CA-125 value from baseline according to GCIG CA-125 criteria
Combined RECIST/CA-125 overall response rate according to GCIG (subjects with ovarian cancer only) | Approximately 2 years
  The proportion of participants with ovarian cancer whose best response is a CR or PR according to the GCIG combined RECIST and CA-125 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne McGoldrick, MD, Study Director — Seagen Inc.
Locations (13):
- United States (7):
  - Women's Cancer Care, Fresno, California
  - Yale Cancer Center, New Haven, Connecticut
  - Florida Cancer Specialists - Lake Nona, Wellington, Florida
  - START Midwest, Grand Rapids, Michigan
  - Oklahoma University at Stephenson Cancer Center, Oklahoma City, Oklahoma
  - START Mountain Region, West Valley City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
- Canada (2):
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - University Health Network, Princess Margaret Hospital, Toronto, Ontario
- START Madrid-CIOCC_Hospital HM Sanchinarro, Madrid, Other, Spain
- Karolinska University Hospital, Stockholm, Other, Sweden
- United Kingdom (2):
  - The Royal Marsden NHS Foundation Trust (RM), London, Other
  - Sarah Cannon Research Institute UK, London, Other